CLINICAL TRIAL: NCT05025553
Title: Gut Mobilization With Oral Administration of Polyethylene Glycol (PEG) at the Dose of 6.9 g/d Once a Day for 6 Months in Chronically Constipated Autistic Children.
Brief Title: Oral Administration of Polyethylene Glycol (PEG) for 6 Months in Chronically Constipated Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Antonio Persico, Full Professor in Child & Adolescent Neuropsychiatry, University of Messina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEG_study_ASD
Record Dates: First submitted 2021-08-15; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Autistic Spectrum Disorder; Constipation
Keywords: Autism; 4-cresol; anxiety; autism spectrum disorder; biomarkers; constipation; microbiota
MeSH Terms: conditions — Autism Spectrum Disorder; Constipation; Autistic Disorder; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: In this open trial, each child underwent gut mobilization using a standard protocol with oral administration of PEG (6.9 g/d once a day) for 6 months. Children were observed and behaviorally tested at baseline (T0), 1 month (T1) and 6 months (T2) after gut mobilization.
  At the time of recruitment, Intellectual Quotient (IQ) or Developmental Quotient (DQ) were determined using the Leiter International Performance Scale-Third Edition or the Griffith Mental Development Scales, respectively. Autistic behaviors were assessed using the ADOS-2, and the Children Autism Rating Scales (CARS). Adaptive functioning was assessed using the Vineland Adaptive Behavior Scales-Second Edition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gut mobilization (Other): Polyethylene Glycol (PEG) at the dose of 6.9 g/d once a day for 6 months.
  Interventions: Dietary Supplement: Gut mobilization

INTERVENTIONS:
Dietary Supplement: Gut mobilization — Polyethylene Glycol (PEG) at the Dose of 6.9 g/d Once a Day for 6 Month. Children were observed and tested at baseline (T0), 1 month (T1) and 6 months (T2) after gut mobilization.

SUMMARY:
Many autistic children suffer from chronic constipation. Gut mobilization was obtained administering polyethylene glycol (PEG) at the dose of 6.9 g/d once a day for 6 months in an open trial involving 21 chronically constipated autistic children 2-8 years old, followed prospectively for 6 months. Children diagnosed with Autism Spectrum Disorder by DSM-5 and confirmed by ADOS-2 criteria, were evaluated before (T0), 1 month (T1), and 6 months (T2) after intestinal mobilization, recording Bristol stool scale scores, urinary p-cresol concentrations, and behavioral scores for social interaction deficits, stereotypic behaviors, anxiety, and hyperactivity.

DETAILED DESCRIPTION:
Chronic constipation is common among children with ASD and is associated with more severe anxiety, hyperactivity, irritability and repetitive behaviors. Young autistic children with chronic constipation display higher urinary and foecal concentrations of p-cresol, an aromatic compound produced by gut bacteria, known to negatively affect brain function. Acute p-cresol administration to BTBR mice enhances anxiety, hyperactivity and stereotypic behaviors, while blunting social interaction. This study was undertaken to prospectively assess the behavioral effects of gut mobilization in young autistic children with chronic constipation, and to verify their correlation with urinary p-cresol. To this aim, 21 chronically constipated autistic children 2-8 years old were evaluated before (T0), 1 month (T1), and 6 months (T2) after intestinal mobilization, recording Bristol stool scale scores, urinary p-cresol concentrations, and behavioral scores for social interaction deficits, stereotypic behaviors, anxiety, and hyperactivity. Gut mobilization was obtained administering PEG (6.9 g/d once a day) for 6 months. A progressive, statistically significant decrease in all behavioral symptoms was recorded over the six-month study period. Urinary p-cresol levels displayed variable trends, mainly increasing at T1 and decreasing at T2. These results support gut mobilization as a simple strategy to at least partly ameliorate ASD symptoms, as well as comorbid anxiety and hyperactivity, in chronically constipated children. These beneficial effects likely involve multiple mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling DSM-5 diagnostic criteria for Autism Spectrum Disorder
* Chronic constipation, namely unsatisfactory defecation characterized by difficult and infrequent passage of lumpy and hard stools during at least the previous 3 months, as reported by parents based on the Bristol Stool Scale

Exclusion Criteria:

* ASD constipated children already treated with laxatives

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change in stool quality | At baseline (T0) prior to gut mobilization; 1 month (T1) and 6 months (T2) after gut mobilization
  Stool quality was assessed by parental report using the Bristol Stool Scale (score ranges from 1 to 7, where 1 is "lumpy constipation" and 7 is "liquid diarrhoea").
Change from baseline urinary concentrations of total p-cresol | First-morning urines were collected at home by parents at baseline (T0), 1 month (T1) and 6 months (T2) after gut mobilization
  Urinary concentrations of total p-cresol, encompassing on average 95% p-cresylsulfate, 3%-4% p-cresylglucuronide and 0.5%-1% of unconjugated free p-cresol, were measured by HPLC three times, averaged and normalized by urinary specific gravity.
Change in Childhood Autism Rating Scale (CARS) | At baseline (T0), 1 month (T1) and 6 months (T2) after gut mobilization
  The Childhood Autism Rating Scale is a clinical rating scale for the trained clinician to rate the presence and severity of signs and symptoms of ASD by direct observation of the child. Scores can range from 15 to 60: below 30, non autistic; 30-36.5 mild to moderate autism; 37-60, severe autism
Change in Repetitive Behavior Scale-Revised (RBS-R) | At baseline (T0), 1 month (T1) and 6 months (T2) after gut mobilization
  44- item questionnaire used to assess repetitive behaviors. Scores range from 0 to 3 (0 = the behavior does not occur, 3 = the behavior is present and severe). Overall rating (last question) ranges from 0 to 100, indicating that the set of behaviors described in the questionnaire do not represent a problem at all (0) or instead represent an extremely severe problem (100).
Change in Conners' Parent Rating Scale - Revised (CPRS-R) | At baseline (T0), 1 month (T1) and 6 months (T2) after gut mobilization
  48-item rating scale used to evaluate through parental reports the presence of childhood hyperactivity/inattention, impulsivity and externalizing behaviors (scores for each item range from 0="not true, never, rarely" to 4="very true, very often or very frequent"; diagnostic threshold score = 60).
Change in Social Responsiveness Scale (SRS) | At baseline (T0), 1 month (T1) and 6 months (T2) after gut mobilization
  65-item questionnaire used to assess social impairment, communication deficits and repetitive behaviors (T scores: <60, normal range; 60-65, mild deficits; 66-75, moderate deficits; 76 or above, severe deficits in reciprocal social behavior).

CONTACTS AND LOCATIONS:
Locations (1):
- Interdipartimental Program "Autismo 0-90" at "G. Martino" University Hospital, Messina, ME, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorrindo P, Williams KC, Lee EB, Walker LS, McGrew SG, Levitt P. Gastrointestinal dysfunction in autism: parental report, clinical evaluation, and associated factors. Autism Res. 2012 Apr;5(2):101-8. doi: 10.1002/aur.237. PMID 22511450
- [Background] Goodhart PJ, DeWolf WE Jr, Kruse LI. Mechanism-based inactivation of dopamine beta-hydroxylase by p-cresol and related alkylphenols. Biochemistry. 1987 May 5;26(9):2576-83. doi: 10.1021/bi00383a025. PMID 3607034
- [Background] Kang DW, Adams JB, Vargason T, Santiago M, Hahn J, Krajmalnik-Brown R. Distinct Fecal and Plasma Metabolites in Children with Autism Spectrum Disorders and Their Modulation after Microbiota Transfer Therapy. mSphere. 2020 Oct 21;5(5):e00314-20. doi: 10.1128/mSphere.00314-20. PMID 33087514
- [Background] Kashyap PC, Marcobal A, Ursell LK, Larauche M, Duboc H, Earle KA, Sonnenburg ED, Ferreyra JA, Higginbottom SK, Million M, Tache Y, Pasricha PJ, Knight R, Farrugia G, Sonnenburg JL. Complex interactions among diet, gastrointestinal transit, and gut microbiota in humanized mice. Gastroenterology. 2013 May;144(5):967-77. doi: 10.1053/j.gastro.2013.01.047. Epub 2013 Feb 1. PMID 23380084
- [Background] Altieri L, Neri C, Sacco R, Curatolo P, Benvenuto A, Muratori F, Santocchi E, Bravaccio C, Lenti C, Saccani M, Rigardetto R, Gandione M, Urbani A, Persico AM. Urinary p-cresol is elevated in small children with severe autism spectrum disorder. Biomarkers. 2011 May;16(3):252-60. doi: 10.3109/1354750X.2010.548010. Epub 2011 Feb 18. PMID 21329489
- [Background] De Angelis M, Piccolo M, Vannini L, Siragusa S, De Giacomo A, Serrazzanetti DI, Cristofori F, Guerzoni ME, Gobbetti M, Francavilla R. Fecal microbiota and metabolome of children with autism and pervasive developmental disorder not otherwise specified. PLoS One. 2013 Oct 9;8(10):e76993. doi: 10.1371/journal.pone.0076993. eCollection 2013. PMID 24130822
- [Background] Gabriele S, Sacco R, Altieri L, Neri C, Urbani A, Bravaccio C, Riccio MP, Iovene MR, Bombace F, De Magistris L, Persico AM. Slow intestinal transit contributes to elevate urinary p-cresol level in Italian autistic children. Autism Res. 2016 Jul;9(7):752-9. doi: 10.1002/aur.1571. Epub 2015 Oct 6. PMID 26437875
- [Background] Gabriele S, Sacco R, Cerullo S, Neri C, Urbani A, Tripi G, Malvy J, Barthelemy C, Bonnet-Brihault F, Persico AM. Urinary p-cresol is elevated in young French children with autism spectrum disorder: a replication study. Biomarkers. 2014 Sep;19(6):463-70. doi: 10.3109/1354750X.2014.936911. Epub 2014 Jul 10. PMID 25010144
- [Background] Pascucci T, Colamartino M, Fiori E, Sacco R, Coviello A, Ventura R, Puglisi-Allegra S, Turriziani L, Persico AM. P-cresol Alters Brain Dopamine Metabolism and Exacerbates Autism-Like Behaviors in the BTBR Mouse. Brain Sci. 2020 Apr 13;10(4):233. doi: 10.3390/brainsci10040233. PMID 32294927
- [Background] Persico AM, Ricciardello A, Lamberti M, Turriziani L, Cucinotta F, Brogna C, Vitiello B, Arango C. The pediatric psychopharmacology of autism spectrum disorder: A systematic review - Part I: The past and the present. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Aug 30;110:110326. doi: 10.1016/j.pnpbp.2021.110326. Epub 2021 Apr 20. PMID 33857522
- [Result] Gevi F, Zolla L, Gabriele S, Persico AM. Urinary metabolomics of young Italian autistic children supports abnormal tryptophan and purine metabolism. Mol Autism. 2016 Nov 24;7:47. doi: 10.1186/s13229-016-0109-5. eCollection 2016. PMID 27904735